CLINICAL TRIAL: NCT06285851
Title: Pilot Study for a Novel Iron-Based Supplement for Athletes
Brief Title: A Novel Iron Supplement for Athletes: Phase I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Lallemand Bio-Ingredients (Other)
Responsible Party: Principal Investigator, Jane Shearer, Principal Investigator, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-0825
Record Dates: First submitted 2024-01-30; First posted 2024-02-29 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Constipation; Diarrhea; Cramp, Abdominal; Bleeding Gastric
MeSH Terms: conditions — Constipation; Diarrhea; Colic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FeSC Cookie (Experimental): Iron-yeast complex
  Interventions: Dietary Supplement: FeSC

INTERVENTIONS:
Dietary Supplement: FeSC — Supplement

SUMMARY:
Female endurance athletes are susceptible to iron deficiency and this can impact their exercise performance. This study is a pilot trial to assess the tolerability of a novel iron supplement prior to conducting a clinical trial on the efficacy of the developed novel iron supplement on iron status and performance.

DETAILED DESCRIPTION:
Current iron supplements on the market are commonly associated with side effects including gastrointestinal distress, nausea, vomiting, and constipation. As a solution, the investigators have developed a novel delivery system for iron supplementation that overcomes many of these limitations. The goal of this study is to assess the tolerability of the developed supplement and any associated symptoms before conducting a clinical trial on this product. Participants will consume 40mg of elemental iron every second day for 14 days. Participants will complete a daily survey in which they will report feelings of stress and recovery as well as gastrointestinal symptoms. Additionally, participants will complete a more thorough survey of gastrointestinal symptoms at baseline, the mid-point, and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* cis-gendered female 18-25years old
* BMI <25 kg/m2
* engaging in moderate to vigorous physical activity for ≥3 hours per week

Exclusion Criteria:

* gastrointestinal issues (e.g. Irritable bowel disease/syndrome)
* chronic illnesses
* prescription medication (including oral contraceptives)
* allergies to supplement ingredients
* iron supplementation in the last 3 months

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
GI Symptoms | Daily for 14 days
  Gastrointestinal Symptoms Questionnaire (rating scale 1-7 where 1= the absence of symptoms and 7=severe symptoms)
Gastrointestinal symptoms | Weekly for 14 days
  Patient-Reported Outcomes Measurement Information System (rating scale 0-4 where 0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much)

SECONDARY OUTCOMES:
Supplement Tolerability and Preferences Questionnaire | 14 days
  Consumer preferences compared to standard of care (rating scale 0-4, where 0=not at all and 4=very much)
Recovery | 14 days
  The Recovery-Stress Questionnaire (rating scale 0-6, where 0=never and 6= always)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Shearer, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaw KA, Tompkins TA, Abrahamson-Durant B, MacNevin G, Parnell JA, MacInnis MJ, Reimer RA, Shearer J. Exploring tolerance and side effects of an innovative yeast-bound iron supplement: a feasibility trial. Pilot Feasibility Stud. 2025 Aug 15;11(1):110. doi: 10.1186/s40814-025-01690-w. PMID 40817080